CLINICAL TRIAL: NCT04411654
Title: An Open-label, Phase 1/2 Study to Evaluate the Safety and Efficacy of Single-dose LY3884961 in Infants With Type 2 Gaucher Disease
Brief Title: Phase 1/2 Clinical Trial of PR001 in Infants With Type 2 Gaucher Disease (PROVIDE)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prevail Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J3Z-MC-OJAB (PRV-GD2-101)
Record Dates: First submitted 2020-05-11; First posted 2020-06-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Gaucher Disease, Type 2
Keywords: Gaucher Disease; GD; Gaucher; Type 2 Gaucher; Neuronopathic Gaucher; nGD; AAV9; GBA; Gene Therapy; Glucocerebrosidase; GBA1 mutation; Infants
MeSH Terms: conditions — Gaucher Disease | interventions — Methylprednisolone; Sirolimus; Prednisone

STUDY DESIGN:
Masking Description: Blinded assessor used in secondary outcome measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose (Experimental)
  Interventions: Genetic: LY3884961; Drug: Methylprednisolone; Drug: Sirolimus; Drug: Prednisone
- High Dose (Experimental)
  Interventions: Genetic: LY3884961; Drug: Methylprednisolone; Drug: Sirolimus; Drug: Prednisone

INTERVENTIONS:
Genetic: LY3884961 — Participants will receive a single dose of LY3884961 administered intracisternally.
Drug: Methylprednisolone — Single IV pulse administered as concomitant medication.
Drug: Sirolimus — Loading dose, followed by maintenance doses, followed by dose tapering; administered as concomitant medication.
Drug: Prednisone — Administered orally as concomitant medication, followed by dose tapering.

SUMMARY:
J3Z-MC-OJAB is an open-label, Phase 1/2, multicenter study to evaluate the safety and efficacy of single-dose LY3884961 (formerly PR001) in infants diagnosed with Type 2 Gaucher disease (GD2). For each patient, the study will be approximately 5 years in duration. During the first 12 months after dosing, patients will be evaluated for the effects of LY3884961 on safety, tolerability, immunogenicity, biomarkers, and efficacy. Patients will be followed up for an additional 4 years to monitor safety and changes on selected biomarkers and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Bi-allelic GBA1 mutations consistent with a diagnosis of GD2 confirmed by the central laboratory.
* Clinical diagnosis of GD2
* Parent/legal guardian is capable of providing signed informed consent; including compliance with the requirements and restrictions listed in the informed consent form (ICF) in this protocol.
* Patient has a parent/legal guardian able to participate in the study as a source of information on the patient's health status and cognitive and functional abilities (including providing input into the rating scales).

Exclusion Criteria:

* Significant CNS disease other than GD2 that may be a cause for the patient's symptoms or interfere with study objectives.
* Achieved independent gait.
* Severe peripheral symptoms of GD which, in the opinion of the Investigator, would pose an unacceptable risk to the patient or interfere with the patient's ability to comply with study procedures or interfere with the conduct of the study.
* Concomitant disease, condition, or treatment which, in the opinion of the Investigator, would pose an unacceptable risk to the patient or interfere with the patient's ability to comply with study procedures or interfere with the conduct of the study.
* Use of any substrate reduction therapy (SRT) for GD treatment.
* Use of prohibited medications, herbals, or over-the-counter agents as listed in the protocol.
* Any type of prior gene or cell therapy.
* Use of systemic immunosuppressant or corticosteroid therapy other than protocol-specified immunosuppression.
* Participation in another investigational drug or device study within the past 3 months.
* Brain MRI (magnetic resonance imaging) and MRA (magnetic resonance angiography) showing clinically significant abnormality deemed a contraindication to intracisternal injection.
* Clinically significant laboratory test result abnormalities assessed at screening.
* Contraindications or intolerance to radiographic visualization methods (e.g. MRI, MRA, CT), and intolerance to contrast agents used for MRI or CT scans.
* Contraindications to general anesthesia or sedation.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Events leading to discontinuation | Year 5
Immunogenicity of AAV9 and GCase in blood | Up to Year 2
Immunogenicity of AAV9 and GCase in CSF | Up to Year 1

SECONDARY OUTCOMES:
Time to death | Baseline until event or study completion, up to Year 5
Time to clinical event | Baseline until event or study completion, up to Year 5
  Clinical event defined as tracheostomy/invasive ventilation, and/or percutaneous endoscopic gastrostomy (PEG) tube placement, and/or nasogastric (NG) tube placement
Change in cognitive function | Months 6,12 and up to Year 2
  Measured using Bayley Scales of Infant and Toddler Development (BSID-III)
Change in cognitive function | Study Month 12 and up to Study Year 2
  Measured using Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV) as appropriate. (Not all patients begin the study at birth. Only patients who are age 36 months at the designated study visits will be assessed using this measure)
Change in motor skills | Months 6, 12 and up to Year 2
  Change from baseline in motor function using Gross Motor Function Measure (GMFM-88).
Change in motor skills | Months 6, 12 and up to Year 2
  Change from baseline in motor function using the BSID-III.
Change in Clinical Global Impressions (Severity) | Months 6, 12 and up to Year 2
  Change from baseline in the clinical severity of illness (CGI-Severity {CGI-S}).
Clinical Global Impressions (Improvement) | Months 6, 12 and up to Year 2
  Clinical improvement from baseline (CGI-Improvement [CGI-I]).
Change in adaptive behavior and functioning | Months 6 and 12 and up to Year 2
  Change from baseline in adaptive functioning using the Vineland Adaptive Behavior Scale (VABS-2) (2nd edition)
Change in most troubling symptoms | Months 6, 12 and up to Year 2
  Change from baseline in the Visual Analog Scale for the Most Troubling Symptoms (VAS-MTS)
Change in behavioral symptoms | Months 6, 12 and up to Year 2
  Change from baseline in the Child Behavior Checklist (CBCL)
Change in GCase (glucocerebrosidase) enzyme activity levels in blood | Up to Year 5
Change in GCase enzyme activity levels in CSF (cerebrospinal fluid) | Up to Year 3
Change in glycolipid levels in blood | Up to Year 5
Change in glycolipid levels in CSF | Up to Year 3
Individual Vector Shedding data | Up to Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Hamzeh Migdadi, M.D., Study Director — Prevail Therapeutics
Locations (5):
- United States (4):
  - UCSF Benioff Children's Hospital, 5700 Martin Luther King Jr Way, Oakland, California
  - University of Minnesota Masonic Children's Hospital, 2450 Riverside Avenue, Minneapolis, Minnesota
  - Children's Hospital of Pittsburgh, 4401 Penn Avenue, Pittsburgh, Pennsylvania
  - Lysosomal & Rare Disorders Research and Treatment Center, Fairfax, Virginia
- Manchester Centre for Genomic Medicine, 6th Floor, St Mary's Hospital, Oxford Road, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No